CLINICAL TRIAL: NCT06815835
Title: A Prospective, Randomized, Parallel, Three-arm, Open-label, Clinical Trial to Evaluate the Immunological Non-interference of Measles and Rubella Vaccine (Live) I.P. (Freeze Dried) of M/s. Zydus Lifesciences Ltd. With Yellow Fever Vaccine Administered to Bangladeshi Healthy Infants Aged 9-12 Months
Brief Title: Non-interference Study of MR and Yellow Fever Vaccines Among Bangladeshi Infants Aged 9-12 Months
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-24098
Record Dates: First submitted 2025-01-22; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Measles; Rubella; Yellow Fever
Keywords: Safety; Non-interference; Measles and Rubella; Co-administration; Immunogenicity
MeSH Terms: conditions — Measles; Rubella; Yellow Fever | interventions — Freeze Drying; Yellow Fever Vaccine

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, parallel, three-arm, open-label, equivalence clinical trial of co-administration of MR vaccines (manufactured by Zydus Lifesciences Limited) and Yellow fever vaccine (WHO prequalified) among healthy infants 9 to 12 months of age in Dhaka, Bangladesh who did not receive any of the aforementioned vaccines will be included in the study.
Masking Description: This is a prospective, randomized, parallel, three-arm, open-label, equivalence clinical trial of co-administration of MR vaccines (manufactured by Zydus Lifesciences Limited) and Yellow fever vaccine (WHO prequalified). The vaccine administration team will be un-blinded to the treatment assignment list. The vaccine administrator team members will not be involved in the evaluation of vaccine safety and laboratory analysis. The DSMB will be responsible for un-blinding the randomization number codes in the event of severe putative vaccine reactions. Otherwise, the codes will not be revealed until the end of the trial and until the computerized dataset has been frozen. If the intervention assignment is un-blinded, all study collaborators will be notified immediately. If deemed necessary, the DSMBs will recommend unblinding to the IRB and contact the study statistician responsible for providing information on the vaccine received by the individual in question.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test (MR+YF) (Experimental): Based on randomization (n= 510) potential participants will be vaccinated with MR+YF on Day 0. A diary card will be provided. A blood sample (4-5 ml) will be collected for immunological assay on Day -1, Week 6 ±3 days, and Week 26 ±7 days. All details will be recorded in the eCRF.
  Interventions: Biological: Measles-Rubella vaccine (Live) I.P. (Freeze Dried) of M/s. Zydus Lifesciences Ltd; Biological: Yellow fever Vaccine (WHO prequalified)
- Reference 1 (MR) (Experimental): Based on randomization (n= 510) potential participants will be vaccinated with MR on Day 0. A diary card will be provided. A blood sample (4-5 ml) will be collected for immunological assay on Day -1, Week 6 ±3 days, and Week 26 ±7 days. All details will be recorded in the eCRF.
  Interventions: Biological: Measles-Rubella vaccine (Live) I.P. (Freeze Dried) of M/s. Zydus Lifesciences Ltd
- Reference 2 (YF) (Placebo Comparator): Based on randomization (n= 510) potential participants will be vaccinated with YF on Day 0. A diary card will be provided. A blood sample (4-5 ml) will be collected for immunological assay on Day -1, Week 6 ±3 days, and Week 26 ±7 days. All details will be recorded in the eCRF.
  Interventions: Biological: Yellow fever Vaccine (WHO prequalified)

INTERVENTIONS:
Biological: Measles-Rubella vaccine (Live) I.P. (Freeze Dried) of M/s. Zydus Lifesciences Ltd — Live attenuated vaccine
  Arms: Reference 1 (MR); Test (MR+YF)
Biological: Yellow fever Vaccine (WHO prequalified) — Live attenuated vaccine
  Arms: Reference 2 (YF); Test (MR+YF)

SUMMARY:
This study will be conducted among 1530 healthy infants of 9 to 12 months of age residing in the Dakshinkhan and Uttarkhan area which is located in Dhaka North City Corporation (DNCC) to enroll the required number of participants. Only infants who have not previously received the MR and YF vaccines will be enrolled. The findings of this study are likely to have a significant impact on vaccine co-administration strategies for campaign and routine immunization programs. The participants will be assigned to one of the three groups by the central computer-generated randomization schedule. The numbers are defined for each arm (Table 1) based on the sample size calculation. A list of infants who did not receive MR and Yellow fever vaccine will be prepared before enrollment by trained study staff (TSS). The TSSs will visit households in the defined study area and ask if the parents/guardians of infants aged 9-12 months are willing to participate in the study. If they show a willingness to participate, the TSSs will check their vaccination cards (if available) and prepare the list of potentially eligible infants who have not received MR and Yellow fever vaccines based on their vaccination card status. The investigators will collect blood specimens (4-5 ml) at the time of screening (visit-1), to evaluate serological markers of dengue and Japanese Encephalitis infection and for baseline (pre-vaccination) immunological assessment. The investigators will vaccinate seronegative, eligible participants within 24 hours of blood collection. There will be additional three follow-up visits after enrollment and will collect around 3-4 ml blood from each participant during visit 4 (week 6), and visit 5 (week 26) for immunological assessment. Diary cards will be used to collect adverse events (AEs) following immunization (AEFI) data for vaccinated participants (up to 14 days for solicited and 6 weeks for unsolicited AEs). Medically attended adverse events (MAAEs) and data on serious adverse events (SAEs) will be reported during the study. All study updates including AEs and SAEs will be reported to the data safety and monitoring board (DSMB) and sponsor.

DETAILED DESCRIPTION:
This is a prospective, randomized, parallel, three-arm, open-label, equivalence clinical trial of co-administration of MR vaccines (manufactured by Zydus Lifesciences Limited) and Yellow fever vaccine (WHO prequalified) among healthy infants 9 to 12 months of age in Dhaka, Bangladesh will be conducted. Infants who did not receive any of the aforementioned vaccines will be included in the study.

Hypothesis:

Seropositivity following concomitant administration of MR and Yellow fever vaccines is equivalent when the vaccines are administered alone

Specific Objectives

Primary objective:

To evaluate the immunological non-interference of co-administration of Measles and Rubella vaccine (Live) I.P. (Freeze Dried) [MR vaccine] of M/s. Zydus Lifesciences Ltd. with Yellow fever [YF] vaccine in healthy infants.

Secondary objective:

To evaluate the safety of co-administration of MR vaccine of M/s. Zydus Lifesciences Ltd. with Yellow fever vaccine in healthy infants.

Study design This will be a prospective, randomized, parallel, three-arm, open-label, equivalence clinical trial to evaluate the immunogenicity and safety of the co-administration of the MR vaccine manufactured by Zydus Lifesciences Ltd. with Yellow fever vaccine in healthy infants aged 9-12 months. The study will be conducted in a population of infants who is residing in a selected geographical catchment area in Dhaka, Bangladesh.

A minimum of 1530 healthy infants aged 9-12 months (age at enrollment, calculated as per completed months) over the study area will be enrolled in this clinical trial to evaluate the immunogenicity and safety of the study vaccines.

Study area Dakshinkhan and Uttarkhan are both located in the Dhaka North City Corporation (DNCC) with distinct population characteristics and geographical areas. Dakshinkhan spans 11 square kilometers and had a population of 416,601 in 2022, resulting in a high population density of 37,872 people per square kilometer. It contains 113,709 households, with an average household size of 3.8 individuals, and a gender distribution of 53.63% male and 46.37% female. In 2023, the birth of 8,884 new children resulted in a birth rate of 21.3 per 1,000 inhabitants. Uttarkhan is larger with an area of 20.5 square kilometers with the population density of 6,153 people per square kilometer, resulting in a total population of 126,149 as of 2022. This population is distributed across 33,901 households, with an average household size of 3.7 individuals. The gender distribution shows 51.91% male and 48.08% female. In 2023, the birth of 2,806 new children in a birth rate of 22.2 per 1,000 inhabitants.

Selection of age-eligible infants by household visit in the study area All households in the study area will be assigned a unique identification number and all household members will be enumerated. Information about the age-eligible infants including name, age, sex, date of birth, and parent's name will be obtained. In addition, the name of the HH head, address, and cell phone number of HHs will be collected. The investigators will take photos of birth certificates or national immunization cards to confirm the age of participants if available. Verbal consent will be provided by either the head of the household or a key informant.

Distribution of participant card for potentially eligible infants for vaccination After preparing the baseline list, the investigators will identify the age-eligible (9-12 months) participants. Then the investigator will prepare participant cards for all eligible infants which will be provided before the vaccination. There will be a unique identification number on the participant card which will be used during vaccination. A master list of potential eligible participants will be prepared.

Informed consent The informed written consent will be presented to the participant's parent/guardian in Bangla detailing no less than the exact nature of the study, what it will involve for the participant, the implications and constraints of the protocol, the known side effects and any risks involved in taking part. It will be clearly stated that the participant's parent/guardian is free to withdraw their child from the study at any time for any reason without prejudice to future care, without affecting their legal rights, and with no obligation to give the reason for withdrawal. The participant and their parents/guardians will be allowed as much time as they wish to consider the information, within the recruitment period, and the opportunity to question the investigator or other independent parties to decide whether they will participate in the study. Written informed consent will then be obtained using the participants' parent/guardian's dated signature or thumbprint and dated signature of the person who presented and obtained the informed consent. The person who obtained the consent must be suitably qualified and experienced and have been authorized to do so by the Principal Investigator (PI). A copy of the signed informed consent will be given to the participant's parents/guardians. The original signed form will be retained at the study site. An impartial witness for the parent/guardian will attest that the information in the consent form and any other written information was accurately explained to, and understood by the parent/guardian and that informed consent was freely given by the parent/guardian. The witness will also sign and date the consent form.

Screening and eligibility assessment Study staff will invite participants to the field office to be enrolled in the study. If agreed, written consent will be obtained from the parent/guardian at the field office. After obtaining informed written consent, the investigators will collect 4-5 ml of blood specimens at the time of screening (visit-1) to evaluate serological markers of dengue infection (NS1 antigen, IgM, and IgG antibodies) and Japanese Encephalitis (IgM and IgG antibodies). The investigators will carry out the aforementioned screening tests because previous studies showed that the prevalence of asymptomatic dengue infections during outbreaks was 59.26%. Most Japanese encephalitis infections are also asymptomatic. So, it is important to conduct screening tests to identify and exclude participants with asymptomatic infections. Additionally, there is a potential for cross-reactivity of Yellow fever antibodies with antibodies generated against other flaviviruses, such as dengue and Japanese encephalitis. Therefore, screening tests are important to exclude participants with pre-existing antibody titres. The remaining blood specimens will be used for baseline (pre-vaccination) immunological assessment. After the screening test, the potentially eligible, seronegative participants will be enrolled for vaccination within 24 hours of blood collection. They will undergo a thorough general physical examination including recording of vitals such as body temperature, heart rate, and respiratory rate. The Participants will be evaluated as per the inclusion and exclusion criteria. Vitals will be recorded and physical examination will be conducted at each follow-up visit and the end of the study visit. After screening, the eligible participant will be enrolled for vaccination in different groups after matching with eligibility criteria. A member of the study team will collect/edit demographic information (including age and address) and participant contact details in the screening case report form (CRF).

Enrollment Potential participants will attend the vaccination site. Upon arrival, inclusion/exclusion criteria will be assessed. The physical examination will be carried out before vaccination. Before vaccination, TSS will ensure that the results of screening tests are available. After completion of the eligibility checking, a sticker will be allocated for the participant which includes the information of vaccination ID and axillary temperature; these will be used in the vaccine accountability log. Based on the randomization of the three groups (mentioned below), the appropriate vaccine will be administered by a trained study staff. The participant will then be vaccinated and will be asked to wait at least 30 minutes for any immediate hypersensitivity reactions or other adverse events (AEs). All details will be recorded in the eCRF (Electronic Case Report Form).

Three Study groups A.Test (MR+YF): MR and YF vaccines administered concomitantly at day 0 B.Reference 1 (MR): MR vaccine administered at day 0 C.Reference 2 (YF): YF vaccine administered at day 0

Randomization The study statistician will prepare computer-generated randomization lists. The enrolled Participants would be assigned to one of the three study groups according to the centralized computer-generated randomization allocation.

Study activities

This study will be conducted as per the methods and procedures described in the visit-wise manner as follows:

Visit 1 / Upto Day -1 (Screening)

* Written informed consent will be taken from the parents or guardians of the participants before performing any study-related activity
* A participant ID number will be assigned once the study-specific consent form has been signed
* Demographic details i.e., age, and gender will be recorded
* Vital signs (body temperature, heart rate, and respiratory rate) will be recorded
* Medical and vaccination history will be obtained and physical examination (length, and weight) will be performed by a physician
* Inclusion/exclusion criteria are reviewed to determine qualification for enrolment.
* Blood specimens (4-5 ml) will be collected for Dengue NS1 antigen, IgM& IgG antibodies and Japanese Encephalitis IgM & IgG antibodies and baseline (pre-vaccination) anti-measles, anti-rubella IgG, and anti-YF antibody titre

Visit 2 / Day 0 (Enrollment, Randomization and Vaccination)

* Clinical evaluation and eligibility criteria will be reviewed by the study physician to evaluate the eligibility for enrollment
* Medical and vaccination history will be recorded
* Vital signs (body temperature, heart rate, and respiratory rate) recording and physical examination will be performed
* Inclusion and exclusion criteria (as mentioned before) will be checked
* Eligible participants will be enrolled
* The participant will be randomized in one of the three study groups as per their allocated randomization number and the allocated study vaccine will be administered
* Assessment of immediate reactions: For group A, the MR vaccine will be administered and the participants will be observed for 30 minutes to monitor for any immediate adverse or anaphylaxis reactions. Then the YF vaccine will be administered and the participants will be observed for another 30 minutes. For groups B and C, the participants will be observed for 30 minutes after each vaccination
* AEs, if any (volunteered by the participants' parents or observed by the investigator/designee) during this observation period will be recorded
* Two diary cards (one for solicited AEs and one for unsolicited AEs) will be provided to participants' parents/guardians to record local (injection site) and systemic AEs. Solicited local AEs will be recorded for 7 days after vaccination, solicited systemic AEs will be recorded for 14 days after vaccination and participants' parents/guardians will be instructed to bring the diary card for solicited AEs at visit 3 (Week 2+3 days). Unsolicited AEs will be recorded for 6 weeks (±3 days) after vaccination. The investigators will collect the diary card for unsolicited AEs at Visit 4 (week 6 ± 3 days). Following visit 4, unsolicited AEs will only be recorded if they are defined as serious adverse events (SAEs) or medically attended adverse events (MAAEs) for 26 weeks (±7 days)

Visit 3 / week 2 + 3 days (Follow-up):

* Vital signs recording and physical examination will be performed
* Medical history including medication will be recorded
* Participants' diary card for solicited AEs will be collected back and reviewed by the investigator/designee
* Solicited AEs, if any, either recorded in the diary card or reported by participants' parents/guardians or observed by the investigator or designee will be recorded

Visit 4/ Week 6 ± 3 days (Follow-up):

* Vital signs recording and physical examination will be performed
* Medical history including medication will be recorded
* Participants' diary card for unsolicited AEs will be collected back and reviewed by the investigator/designee
* Unsolicited AEs, if any, reported by participants' parents/guardians, or observed by the investigator or designee will be recorded
* A 3-4 ml blood sample will be collected for assessment of post-vaccination anti-measles, anti-rubella IgG, and anti-YF antibody titre

Visit 5 / Week 26 ± 7 days (End of study):

* Vital signs recording and physical examination will be performed
* Medical history including medication will be recorded
* MAAEs, if any, will be recorded
* A 3-4 ml blood sample will be collected to assess post-vaccination anti-measles, anti-rubella IgG, and anti-YF antibody titre

Investigational Medicinal Product (IMP)

Measles-Rubella vaccine (Live) I.P. (Freeze Dried) of M/s. Zydus Lifesciences Ltd.

* The vaccine will be available in 5-dose presentation in lyophilized form and will be reconstituted with the diluent supplied along with the vaccine immediately prior to vaccination. Each single dose of 0.5 ml after reconstitution contains not less than 1000 CCID50 Live Attenuated Measles Virus (Edmonston Zagreb Strain) propagated on human diploid cells, and 1000 CCID50 Live Attenuated Rubella Virus (RA 27/3 Strain) propagated on Human Diploid Cells
* The reconstituted 0.5 ml single dose of the vaccine will be administered as a subcutaneous injection in the anterolateral aspect of the upper thigh taking care of aseptic precautions.
* Each vial of test vaccine will be used for a single participant
* The remaining 2.0 ml of unused reconstituted vaccine will be kept for accountability and must not be used for vaccination of any other participant

Yellow fever Vaccine (WHO prequalified)

* The vaccine will be available as either a single-dose or multi-dose presentation in lyophilized form and will be reconstituted with the diluent supplied along with the vaccine immediately prior to vaccination
* The reconstituted 0.5 ml single dose (SD) of the vaccine will be administered as a subcutaneous injection in the anterolateral aspect of the upper thigh taking care of aseptic precautions
* If a multi-dose presentation of the vaccine is used then the remaining unused reconstituted vaccine will be kept for accountability and it must not be used for the vaccination of any other participant In the test group, both MR and YF vaccines will be administered concomitantly as separate injections in different thighs.

Supply The test and reference vaccines will be provided by Zydus Lifesciences Limited.

Storage The study vaccines (both the lyophilized and reconstituted vaccines) will be stored in the dark at a temperature between 2º-8º C in temperature-monitored icddr,b cold room facilities, when not in use for daily activities. The vaccines will be stored in temperature-monitored refrigerators or cool boxes, when in use for daily activities. The diluent should not be frozen but should be kept cool.

Each vial of the MR vaccine will be labelled with a "vaccine vial monitor" (VVM); a temperature-sensitive dot that provides an indication of the cumulative heat to which the vial has been exposed. It warns the end-user when exposure to heat is likely to have degraded the vaccine beyond an acceptable level and should not be used.

Special precautions for storage

* Store at 2°C to 8°C
* Do not freeze. Discard if frozen.
* Shake gently before use.
* Do not use the vaccine after the expiration date shown on the label

Accountability of the Study Vaccine The vaccines will be shipped to a central storage facility in Bangladesh and passed through customs. It will then be transported and distributed to local vaccination sites while maintaining the cold chain (aiming for a temperature between 2º-8ºC). The number of doses of study vaccines that are received, used, and wasted will be documented daily during the study and checked weekly.

Adverse events After administration of the study vaccine, participants will be observed closely for at least 30 minutes for any immediate hypersensitivity reactions or any other adverse events (AEs). All details will be recorded in the CRF. Two diary cards will be given to each participant on the day of vaccination. Parents of participants will be encouraged to go to the 'adverse event monitoring cell' at the Dakshinkhan field office which will have a medical doctor and also available on-call 24 hours a day for adverse event monitoring throughout the whole vaccination period.

Procedures to Evaluate an Adverse Event Definitions Adverse Event following immunization (AEFI): Any untoward medical occurrence which follows immunization and which does not necessarily have a causal relationship with the usage of the vaccine. The adverse event may be any unfavourable or unintended sign, abnormal laboratory finding, symptom or disease.

Serious Adverse Events (SAEs):

Any untoward medical occurrence at any dose:

1. Results in death,
2. Is life-threatening,
3. Requires inpatient hospitalization or prolongation of existing hospitalization,
4. Results in persistent or significant disability/incapacity,
5. Is a congenital anomaly/birth defect
6. Requires intervention to prevent permanent impairment or damage.

Medically Attended Adverse Events (MAAEs): MAAEs are defined as AEs with medically attended visits including hospital, emergency room, or other visits to or from medical personnel for any reason. Adverse events (e.g., abnormal vitals) identified at a routine study visit will not be considered MAAEs.

Adverse Events Recording After administration of the study vaccine(s), participants will be observed closely for at least 30 minutes for any immediate hypersensitivity reactions or any other adverse events (AEs).

Diary card - Test group (MR+YF) After concomitant administration of MR and YF vaccines, the participants' parents will be provided two diary cards to record solicited and unsolicited AEs that may occur after vaccination. Solicited local AEs (pain, redness, swelling, and induration) will be recorded for 7 days after vaccination; and solicited systemic AEs (fever, rashes, running nose, cough, diarrhea, vomiting, abnormal crying, loss of appetite, drowsiness and irritability) will be recorded for 14 days after vaccination. Unsolicited (other) AEs will be recorded for 6 weeks post-vaccination. The diary cards will be collected during the follow-up visits after 14 days (solicited AEs) and 6 weeks (unsolicited AEs) post-vaccination.

Diary card - Reference 1 group (MR) After administration of the MR vaccine, the participants' parents will be provided with two diary cards to record solicited and unsolicited AEs that may occur after vaccination. Solicited local AEs (pain, redness, swelling, and induration) will be recorded for 7 days after vaccination; and solicited systemic AEs (fever, rashes, running nose, cough, diarrhea, vomiting, abnormal crying, loss of appetite, drowsiness and irritability) will be recorded for 14 days after vaccination. Unsolicited (other) AEs will be recorded for 6 weeks. The diary cards will be collected during the follow-up visits after 14 days (solicited AEs) and 6 weeks (unsolicited AEs) post-vaccination.

Diary card - Reference 2 group (YF) After administration of the YF vaccine, the participants' parents will be provided two diary cards to record solicited and unsolicited AEs that may occur after vaccination. Solicited local AEs (pain, redness, swelling & induration) will be recorded for 7 days after vaccination; and solicited systemic AEs (fever, rashes, vomiting, abnormal crying, loss of appetite, drowsiness and irritability) will be recorded for 14 days after vaccination. Unsolicited (other) AEs will be recorded for 6 weeks. The diary card will be collected during the follow-up visits after 14 days (solicited AEs) and 6 weeks (unsolicited AEs) post-vaccination.

After 6 weeks post-vaccination, unsolicited AEs will only be recorded if they are defined as serious adverse events (SAEs) or medically attended adverse events (MAAEs).

Follow-up of AE, even after the date of study completion, is required if the AE or its sequelae persist. Follow-up is required until the event or its sequel resolves or stabilizes at a level acceptable to the investigator.

All the AEs will be documented in the respective CRFs including Type of AE, Date of onset, Severity, Treatment given, Association or relationship to the study vaccine, Date of resolution, Duration, Outcome, Whether the AE is serious or not

Additionally, if any participants present with symptoms of rubella or measles during the study follow-up visit, diagnostic tests will be conducted for further management.

Discontinuation of the Study due to Adverse Events:

The reason for a participant discontinued from the study will be recorded in the CRF. Discontinuation occurs when an enrolled participant ceases participation in the study, regardless of the circumstances, before the completion of the study. Discontinuation must be reported immediately to the sponsor if it is due to the SAE. The final evaluation as required by the Protocol will be performed at the time of discontinuation if medically acceptable or as soon as possible after that. The Investigator will record the reason for study discontinuation and, if possible, provide or arrange for appropriate follow-up and document the cause of the participant's condition.

Causality assessment of adverse events:

Causality (relatedness) of AE to the study vaccine will be assessed by the Investigator as per the following categories:

* Related: There is suspicion that there is a relationship between the study vaccine and the AE (without determining the extent of probability); there is a reasonable possibility that the study vaccine contributed to the AE
* Not Related: There is no suspicion that there is a relationship between the study vaccine and the AE; there are other more likely causes and administration of the study vaccine is not suspected to have contributed to the AE

Unsolicited adverse events:

The AEs other than those listed under the solicited AEs will be considered as unsolicited AEs. Moreover, the AEs listed under solicited local AEs but reported after 7 days post-vaccination or AEs listed under solicited systemic AEs but reported after 14 days post-vaccination will also be considered as unsolicited AEs (i.e., the onset of injection site swelling 7 days after vaccination, the onset of fever 14 days after vaccination, etc.)

All unsolicited AEs occurring within 6 weeks post-vaccination will be recorded. After 6 weeks post-vaccination, unsolicited AEs will only be recorded if they are defined as serious adverse events (SAEs) or medically attended adverse events (MAAEs). The grading of unsolicited AEs, will be assessed as per the following table.

All solicited and unsolicited AEs as mentioned above, regardless of treatment group or suspected causal relationship to the study vaccines will be recorded on the AE page of the CRF. Safety data including adverse events will be tabulated for clinical review.

Serious Adverse Events (SAEs) Serious Adverse Events (SAEs), as judged by a medically qualified investigator, observed by the investigator, or members of the study team, or reported by the parent, will be recorded on the CRF.The following information will be recorded: description, date of onset and end date, severity, assessment of relatedness to study medication, and action taken. Follow-up information should be provided as necessary. All SAEs will be recorded in the CRFs, for the entire study duration. Participants with SAEs will be followed by a medically qualified investigator either until resolution or the event is considered stable.

Reporting procedures for serious adverse events The forms developed by the icddr,b institutional review board (IRB) will be used for reporting all SAEs.

All SAEs occurring within the 6 months post-vaccine administration will be reported to the Data Safety Monitoring Board (DSMB), Directorate General of Drug Administration (DGDA), the PI, and the other study investigators within 24 hours of the site study team becoming aware of the event. The initial reporting will be done by PI only. A more detailed report form will be completed and sent within the shortest period (but not later than 7 days) of the initial report, to all parties mentioned above. Additional and further requested information (follow-up or corrections to the original case) will be detailed in subsequent safety report forms. All SAEs must be reported to the study sponsor within 2 days. Summary reports will be submitted to the icddr,b IRB, and DGDA at the end of the study.

Safety monitoring committee A DSMB will also be formed to oversee the safety component of the study. The DSMB members will not be involved in the study in any way. In addition, a physician with relevant study-related or therapeutic expertise will be identified as an independent safety monitor (ISM). The ISM will not be an investigator for this study. Under any circumstances, the identified ISM would be requested to carry out an independent assessment of the child presented with adverse events. The assessment details will be reported to the PI and DSMB.

Concomitant medication Medications considered necessary for the participants and which will not interfere with the study vaccine may be allowed at the discretion of the principal investigator. Drugs that may interact with the study vaccine will not be permitted during the study period.

* Appropriate records of the same will be kept in the CRF
* A list of all the concomitant medications consumed by the participants would be recorded in the CRF.

Prohibited therapies

The following therapies will be considered as prohibited for vaccinees:

* Any other vaccine administration will be prohibited for 4 weeks after the study vaccine administration
* Aspirin (acetylsalicylic acid) will be prohibited for 4 weeks after the study vaccine administration
* Anti-coagulants will be prohibited within 7 days of the study vaccine administration
* Immunosuppressive agents, immunostimulant agents, immunoglobulins, blood or blood products will be prohibited for the entire study period

Laboratory procedure

Immunogenicity assessment A total of 10-13 ml blood sample will be collected three times in the study; during visit 1 / day -1 (prior to vaccination), visit 4 / week 6, and visit 5 / week 26 for assessment of serum anti-measles, anti-rubella IgG (Immunoglobulin G) and anti-YF antibodies. Upon collection, the blood samples will be stored in cool boxes maintaining a temperature of 2°C-8°C. It will then be transported to the laboratory maintaining a temperature of 2°C-8°C to ensure sample integrity. Once at the lab, the samples will be centrifuged to separate the serum. The serum will then be divided into three approximately equal aliquots and stored at -80°C. One aliquot will be used for the immunogenicity assessment of serum anti-measles and anti-rubella IgG antibodies, utilizing commercial NovaLisa® ELISA kits from NovaTec Immundiagnostica GmbH, Germany, or other available commercial kits. The cut-off titres for evaluating seropositivity and seroconversion rates will be considered as defined in the kit literature. The other aliquot will be sent to the sponsor (Zydus Lifesciences Ltd) or the sponsor's designated reference laboratory for detection of neutralizing antibodies, a reliable correlate of protection induced by YF vaccination, by the Plaque Reduction Neutralization Test (PRNT). The YF virus is a Risk Group 3 pathogen in the WHO and European classification. Also, all biological specimens should be considered potentially infectious and specimens should be handled in a Biosafety Level 3 (BSL3) laboratory. Therefore, the investigators plan to ship the specimens abroad to carry out the PRNT assay in a reference laboratory. A separate manual/working instruction will be prepared to define the procedures for blood sampling and its processing, serum sample storage and transport, etc.

Withdrawal of participants

Participants' parents/guardians can withdraw consent at any point. The investigator may also discontinue a participant from the study at any time if the investigator considers it necessary for any reason including:

* Ineligibility (either arising during the study or retrospectively having been overlooked at screening)
* Significant protocol deviation
* Significant non-compliance with treatment regimen or study requirements
* An adverse event or disease progression resulting in the inability to continue to comply with study procedures and follow-up

Depending on which aspects participants wish to withdraw from, the withdrawal will result in the cessation of any follow-up calls, visits, or blood tests (as applicable to the subset). No further treatment is required in the study, so no additional action will need to take place. Participants' parents/guardians will have the choice when withdrawing, to withdraw from active study procedures only (follow-up calls and visits) but allow us to access their hospital records and blood test results, or withdraw from all study contact. Data and blood samples collected prior to the time of participant withdrawal will be kept and analyzed as part of the study data. A participant who withdraws from the study has the option to re-engage at a future date if they choose to do so. All participants who withdraw from the study will be given information on how to re-engage with the study if they so choose. Reasons for withdrawal from the study, if known, will be recorded in the participant's CRF.

Data management The investigators will populate the content of participants' CRFs and all the study data will be recorded directly into an Electronic Data Capture (EDC) system (Octalsoft). Electronic devices and hard copies of CRFs will be used to collect and record data. Data will be collected online and uploaded to a cloud server regularly when electronic devices are brought back to the central field office, and reliable internet is available. Paper CRFs (pCRFs) will also be available as backup, in case of interruption of online data collection, pCRFs will be used for collecting data and data will then be entered into the EDC system when feasible.

Sample Size Calculation and Outcome The number and percentage of seropositivity rates who exhibit at least 9 NovaTec Units (NTU) for anti-measles antibodies titer to the study participants will be compared between the study groups (Test vs. reference1 and Test vs. reference2). Equivalence will be confirmed if the lower limit and upper limit of two-tailed 95% CI of the difference of seropositivity rate between the Test vaccine and Reference vaccine groups within the margin of ±10%. Considering the above assumptions and a minimum of 70% seropositivity rate with a 10% attrition rate and 90% study power, the investigator has to enroll a total of 1530 healthy participants in this study with 1:1:1 allocation in the study groups (Test - 510; Reference 1 - 510; Reference 2 - 510).

ELIGIBILITY:
Inclusion Criteria:

* The participant must satisfy all the following criteria to be eligible for enrolment:
* Healthy infant participants of either gender aged* 9 to 12 months at the time of enrollment
* Participants should be in good health as determined by the medical history and physical examination based on the clinical judgment of the investigator
* No previous history of vaccination against measles, rubella, or Yellow fever
* Written informed consent from the participant's parent/guardian
* Participant's parent/guardian literate enough to fill the diary card *Age calculated as per completed month

Exclusion Criteria:

* Participants positive for serological markers against Dengue and/or Japanese Encephalitis infections
* History of hypersensitivity reaction to any component of the study vaccines including egg and chicken proteins
* History of hypersensitivity reaction to neomycin
* History of laboratory-confirmed or suspected measles, rubella, or Yellow fever in the past
* Participant exposed# to measles, rubella, or Yellow fever virus within the past 30 days
* Fever of any origin or infectious disorder of 3 days or more within the past month
* Febrile illness (axillary temperature ≥37.5°C) at the time of enrollment
* History of any vaccination within the past month
* Clinically significant systemic disorders such as cardiovascular, respiratory, neurologic, gastrointestinal, hepatic, renal, endocrine, haematological, immunological, or metabolic disorder
* Confirmed or suspected immunosuppressive or immunodeficiency disorder; or participants on any immunosuppressive or immunostimulant therapy
* Known case of thrombocytopenia or any coagulation disorder, or participants on anticoagulation therapy
* Participants administered blood, blood-containing products, or immunoglobulins within the last 3 months or planned administration during the study
* Participant participated in another clinical study in the past 3 months
* Any other reason for which the investigator feels that the participant should not participate #Close contact (family member or neighbour) with laboratory-confirmed or clinical diagnosis of measles/rubella/Yellow fever

Ages: 9 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1530 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Seropositivity | 06 weeks
  Equivalence for seropositivity rate for anti-measles, anti-rubella, and anti-YF IgG antibodies at 6 weeks post-vaccination

SECONDARY OUTCOMES:
Immunogenicity | 06 months
  * Seropositivity rate for anti-measles (≥9 NovaTec Units), anti-rubella (≥10 IU/ml), and anti-YF IgG (Plaque Reduction Neutralization Test titre of ≥1:10) antibodies at 26 weeks post-vaccination
  * Seroconversion rate for anti-measles (≥9 NovaTec Units), anti-rubella (≥10 IU/ml), and anti-YF IgG (Plaque Reduction Neutralization Test titre of ≥1:10) antibodies at 6 weeks and 26 weeks post-vaccination
  * Geometric mean titre of anti-measles, anti-rubella, and anti-YF IgG antibodies at 6 weeks and 26 weeks after vaccination
Safety reporting | 06 months
  * Number of solicited local and systemic adverse events reported during the study
  * Number of unsolicited adverse events reported during the study
  * Number of medically attended adverse events reported during the study
  * Number of serious adverse events reported during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Icddr,B, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cracknell Daniels B, Gaythorpe K, Imai N, Dorigatti I. Yellow fever in Asia-a risk analysis. J Travel Med. 2021 Apr 14;28(3):taab015. doi: 10.1093/jtm/taab015. PMID 33506250
- [Background] Sacchetto L, Drumond BP, Han BA, Nogueira ML, Vasilakis N. Re-emergence of yellow fever in the neotropics - quo vadis? Emerg Top Life Sci. 2020 Dec 11;4(4):399-410. doi: 10.1042/ETLS20200187. PMID 33258924
- [Background] Roukens AH, Visser LG. Yellow fever vaccine: past, present and future. Expert Opin Biol Ther. 2008 Nov;8(11):1787-95. doi: 10.1517/14712598.8.11.1787. PMID 18847312
- [Background] Monath TP, Vasconcelos PF. Yellow fever. J Clin Virol. 2015 Mar;64:160-73. doi: 10.1016/j.jcv.2014.08.030. Epub 2014 Oct 24. PMID 25453327
- [Background] Gaythorpe KA, Hamlet A, Jean K, Garkauskas Ramos D, Cibrelus L, Garske T, Ferguson N. The global burden of yellow fever. Elife. 2021 Mar 16;10:e64670. doi: 10.7554/eLife.64670. PMID 33722340
- [Background] Monath TP. Yellow fever vaccine. Expert Rev Vaccines. 2005 Aug;4(4):553-74. doi: 10.1586/14760584.4.4.553. PMID 16117712
- [Background] Asish PR, Dasgupta S, Rachel G, Bagepally BS, Girish Kumar CP. Global prevalence of asymptomatic dengue infections - a systematic review and meta-analysis. Int J Infect Dis. 2023 Sep;134:292-298. doi: 10.1016/j.ijid.2023.07.010. Epub 2023 Jul 16. PMID 37463631
- [Background] Turtle L, Solomon T. Japanese encephalitis - the prospects for new treatments. Nat Rev Neurol. 2018 Apr 26;14(5):298-313. doi: 10.1038/nrneurol.2018.30. PMID 29697099
- [Background] Endale A, Medhin G, Darfiro K, Kebede N, Legesse M. Magnitude of Antibody Cross-Reactivity in Medically Important Mosquito-Borne Flaviviruses: A Systematic Review. Infect Drug Resist. 2021 Oct 19;14:4291-4299. doi: 10.2147/IDR.S336351. eCollection 2021. PMID 34703255
- [Background] Shi N, Rasuli A, Thollot Y. Safety of two doses of an inactivated hepatitis a vaccine given 6 months apart in healthy toddlers, children, and adolescents aged 12 months to 15 years in China: a phase IV study. Hum Vaccin Immunother. 2019;15(3):748-754. doi: 10.1080/21645515.2018.1539600. Epub 2018 Dec 5. PMID 30403910
- [Background] Nolan T, McVernon J, Skeljo M, Richmond P, Wadia U, Lambert S, Nissen M, Marshall H, Booy R, Heron L, Hartel G, Lai M, Basser R, Gittleson C, Greenberg M. Immunogenicity of a monovalent 2009 influenza A(H1N1) vaccine in infants and children: a randomized trial. JAMA. 2010 Jan 6;303(1):37-46. doi: 10.1001/jama.2009.1911. Epub 2009 Dec 21. PMID 20026597
- [Background] Brandriss MW, Schlesinger JJ, Walsh EE, Briselli M. Lethal 17D yellow fever encephalitis in mice. I. Passive protection by monoclonal antibodies to the envelope proteins of 17D yellow fever and dengue 2 viruses. J Gen Virol. 1986 Feb;67 ( Pt 2):229-34. doi: 10.1099/0022-1317-67-2-229. PMID 3944585
- [Background] Monath TP. Yellow fever: an update. Lancet Infect Dis. 2001 Aug;1(1):11-20. doi: 10.1016/S1473-3099(01)00016-0. PMID 11871403
- [Background] Measles vaccines: WHO position paper - April 2017. Wkly Epidemiol Rec. 2017 Apr 28;92(17):205-27. No abstract available. English, French. PMID 28459148
- See also: WHO. Rubella vaccines: WHO position paper. Wkly Epidemiol Rec. WHO: WHO; 2020 — https://www.who.int/publications/i/item/WHO-WER9527
- See also: Organization CDSC. Summary of product characteristics Measles and Rubella Vaccine (Live) I.P. (Freeze Dried) 2024 — https://www.cdsco.gov.in/opencms/resources/UploadCDSCOWeb/2018/UploadSmPC/R%20Vaccine%20Biological%20E.pdf
- See also: WHO. Yellow fever: WHO; 2023 [updated 31 May 2023 — https://www.who.int/news-room/fact-sheets/detail/yellow-fever
- See also: WHO. Yellow Fever Vaccines WHO web page: WHO — https://www.who.int/teams/immunization-vaccines-and-biologicals/diseases/yellow-fever
- See also: WHO. Laboratory biosafety manual, 3rd edition. 2004 — https://www.who.int/publications/i/item/9241546506
- See also: Union E. Directive 2000/54/EC of the European Parliament and of the Council of 18 September 2000 on the protection of workers from risks related to exposure to biological agents at work (seventh individual directive within the meaning of Article 16(1) of — https://eur-lex.europa.eu/eli/dir/2000/54/oj/eng